CLINICAL TRIAL: NCT02945501
Title: Transcranial Electrical Stimulation at Slow Oscillation Frequency During NREM Sleep: An Assessment of Effects on the Restorative Properties of Sleep
Brief Title: Transcranial Electrical Stimulation (TES) at Slow Oscillation (SO) Frequency During NREM Sleep
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Collaborators: Walter Reed Army Institute of Research (WRAIR) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: WRAIR 2262; S-16-11 (Other: Sponsor); USAMRDC (Other: Sponsor)
Record Dates: First submitted 2016-10-21; First posted 2016-10-26 (Estimated); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Sleep Deprivation; Mental Competency
MeSH Terms: conditions — Sleep Deprivation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Subjects Who Received TES SO (Experimental): Participants will sleep for approximately a two hour period and receive TES SO via the NeuroConn DC Stimulator PLUS during the second hour of that two hour sleep period. They will then experience a 46 hour period of sleep deprivation, during which cognitive performance, mood and subjective and objective aspects of sleepiness will be assessed approximately every 75 minutes beginning on the night of restricted sleep/treatment.
  Interventions: Device: NeuroConn DC Stimulator PLUS
- Received SHAM (no TES SO) (Sham Comparator): Participants will sleep for approximately a two hour period and receive a SHAM (no TES SO) during the second hour of that two hour sleep period. They will then experience a 46 hour period of sleep deprivation, during which cognitive performance, mood and subjective and objective aspects of sleepiness will be assessed approximately every 75 minutes beginning on the night of restricted sleep/treatment.
  Interventions: Device: SHAM TES

INTERVENTIONS:
Device: NeuroConn DC Stimulator PLUS — Prior to bedtime on the sleep restriction night, 4 transcranial stimulation electrodes (two on each hemisphere) will be applied to the scalps of each subject. Subjects will receive a one hour period of SO stimulation, for a total of approximately two hours of sleep.
  Arms: Subjects Who Received TES SO
Device: SHAM TES — Prior to bedtime on the sleep restriction night, 4 placebo transcranial stimulation electrodes (two on each hemisphere) will be applied to the scalps of each subject. Subjects will sleep for approximately 2 hours without stimulation.
  Other Names: Placebo
  Arms: Received SHAM (no TES SO)

SUMMARY:
The purpose of this study is to determine if the enhancement of electroencephalographic (EEG) slow-wave activity using transcranial electrical stimulation (TES) at Slow Oscillation (SO) frequency, during a restricted period of nocturnal sleep, enhances the restorative properties of that period of sleep and improves performance during a subsequent period of sleep deprivation.

DETAILED DESCRIPTION:
40 subjects will be enrolled and randomized to participate in this study. A 60 minute TES stimulation sequence consisting of a SO frequency stimulation (TES SO) using the NeuroConn DC Stimulator PLUS or a sham stimulation will be administered during the second hour of a two hour nocturnal sleep period. During wake period subjects will be tested using various cognitive, subjective and objective sleepiness and mood measures. Vital signs measurements will be taken to monitor general health issues. Up to 4 subjects will be enrolled per study session. Due to logistical reasons, no more then 2 subjects per session can be assigned to the TES SO group.

Screening visit = approx. 2 hours At-home component = 7 days In-laboratory study period = 138 hours Total in-laboratory period = approx. 138 hours per subject Total participation time (at home + in-laboratory components) = 15 days

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and non-pregnant, non-lactating women 18 to 39 years of age (inclusive)
* Must demonstrate adequate comprehension of the protocol, by achieving a score of at least 80% correct on a short multiple-choice quiz. Individuals who fail to achieve a passing score on the initial quiz will be given one opportunity to retest after a review of protocol information. Individuals who fail the comprehension assessment for the second time will be disqualified.

Exclusion Criteria:

* Self-reported habitual nightly sleep amounts outside the target range of 6 - 9 hours (i.e., less than 6 hours per night or more than 9 hours per night, on average) (Post-consent Checklist)
* Self-reported nighttime lights-out times earlier than 2100 hours on average during weeknights (Sunday through Thursday) or later than 2300. (Post-consent Checklist)
* Self-reported morning wake-up times later than 0800 on average during weekdays (Monday through Friday) (Post-consent Checklist)
* Self-reported habitual napping (> 1 time a week in conjunction with normal sleep habits) (Post-consent Checklist)
* A rating of 6 or below on question 2 or 3 of the Nonrestorative Sleep Scale, indicating the subject experiences relatively non-refreshing sleep
* An average time to sleep onset of greater than 20 minutes as indicated on the Post-consent Checklist
* Self-reported caffeine use in excess of 400 mg (e.g., approximately 8 caffeinated sodas or 4 12-oz cups of coffee) per day on average (Post-consent Checklist; document provides exclusionary limits for various caffeinated products).
* Score of lower than 31 or higher than 69 on the Morningness-Eveningness Questionnaire (MEQ form)
* Score of 14 or above on the Beck Inventory Form (BDI form)
* Score of 41 or above on the Self-Evaluation Questionnaire
* History of cardiovascular disease (to include but not limited to arrhythmias, valvular heart disease, congestive heart failure, history of sudden cardiac death or myocardial infarction) (Medical History and Examination Form)
* History of neurologic disorder (to include, but not limited to epilepsy or another seizure disorder, amnesia for any reason, hydrocephalus, MS, narcolepsy or other sleep disorders) (Medical History and Examination form; sleep items on Post-Consent Checklist)
* Underlying pulmonary disease requiring daily inhaler use (Medical History and Examination form)
* Kidney disease or kidney abnormalities (Medical History and Examination form, laboratory results)
* Liver disease or liver abnormalities (Medical History and Examination form, laboratory results)
* Self-reported history of psychiatric disorder requiring hospitalization or psychiatric product within the last 2 years or for more than 3 months at one time. (Medical History and Examination form)
* Self-reported or suspected regular nicotine use or addiction, defined as more than 1 cigarette or equivalent per week, within the last 1 year (Medical History and Examination form)
* Self-reported or suspected heavy alcohol use; minimum limit to define heavy alcohol use is 14 drinks per week or as determined by the examining appropriately licensed study investigator (Medical History and Examination form)
* Self-reported or suspected use of products or drugs that cannot be safely discontinued during in-laboratory phases, to be determined on a case-by-case basis by the examining appropriately licensed study investigator (Medical History and Examination form)
* Self-reported or suspected current use of other illicit drugs, to include but not limited to benzodiazepines, amphetamines, cocaine, marijuana (Medical History and Examination form)
* Positive urine pregnancy result
* Resting blood pressure above 140/90 or resting pulse > 110 (Medical History and Examination form). Note that if a repeat measurement is within range then the volunteer will not be excluded.
* BMI ≥ 30 (Obese Class I or greater) (Medical History and Examination form)
* Clinically significant values (as determined by the appropriately licensed study investigator reviewing the study) for any hematology or chemistry parameter. The appropriately licensed study investigator reviewing the laboratory values may opt to repeat any clinically significant tests and include volunteers whose repeat test values are not clinically significant.
* Positive urine nicotine/cotinine result during screening visit (NicCheck™ I test strip results)
* Positive urine drug result during screening visit
* Any use of sleep aids during the 1 year prior to screening
* Inability to read and sign consent
* Lack of access to a quiet, dark environment conducive to sleep from 2100 until 0700 during a seven night period at the beginning of the study
* Participation in any ongoing clinical trials.
* The preceding exclusionary criteria are known to alter sleep (e.g., epilepsy; some neurological disorders), substantially increase inter-subject variability, and/or the disease or condition puts the subject outside the range of what is considered healthy. The PI also maintains the prerogative to disqualify a volunteer if it is deemed that the volunteer's participation would be unsafe for the volunteer or staff or would be disruptive to study conduct or their inclusion could compromise data integrity.
* Volunteers meeting the Beck cut-off (a score of at least 14) and who carry health insurance will be instructed to call their health insurance Mental Health / Substance Abuse referral number.
* Volunteers meeting the first cut-off (score of at least 14 who are not insured will be provided with a community mental health referral contact specific to their county of residence.
* The review of the medical history with the volunteer and the physical examination itself will be performed by an appropriately licensed study investigator. Results of screening urine and blood tests will be reviewed by an appropriately licensed study investigator. The Post-consent Checklist will be administered by a trained research technician and reviewed by the study principal investigator or an appropriately licensed study investigator. If an appropriately licensed study investigator deems it medically advisable, the investigator will share abnormal results with the volunteer, who will be referred to his/her personal physician for follow-up.
* A volunteer who has been cleared for participation may participate in a session if the first day of the session is within 90 days of the screening date. If the first day of the study session is 91 or more days since the volunteer has been screened, the volunteer must re-screen to ensure there has not been a change in eligibility status.

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-10-27 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Point of care safety | Change from baseline at Days 8 - 15. Assessments will be conducted twice a day throughout all wakeful portions of in-laboratory period of study
  Number of Participants With Abnormal Laboratory Values and/or Adverse Events That Are Related to Treatment. Vital signs (blood pressure, pulse, and temperature) will be recorded and abnormal values will be reported to PI who will determine if events meet criteria and definition of an unanticipated device effect (UADE).

SECONDARY OUTCOMES:
Measure the effects of sleep deprivation/sleep restriction on performance using the Psychomotor Vigilance Task (PVT) | Days 11, 12, 13, 14 and 15
  Performed at approximately 75 minutes intervals throughout the waking period, beginning approximately one hour post-awakening on the day prior to sleep restriction and on the recovery day and on night of sleep restriction.
Measure the efficiency and accuracy of simple arithmetic processing using the Mathematical Processing Subtest of the Automated Neuropsychological Assessment Metrics 4 (ANAM4) | Performed at approximately 75 minute intervals throughout waking period, beginning approximately one hour post-awakening on the day prior to sleep restriction and on the recovery day. Days 11 - 15
  Computer based series of mathematical calculations consisting of 3 single digit numbers (e.g. 3+4-5) and indicate if the value of the answer is less than or greater than 5.
Measure current mood states using the Mood Analogue Scale (MAS) | Performed at approximately 75 minute intervals (+/-10 minutes) throughout the waking period, beginning approximately one hour post-awakening on the day prior to sleep restriction and on the recovery day and on the night of sleep restriction. Days 11 - 15
  Computer based self adjective checklist to measure mood states along six subscales: tension-anxiety, anger-hostility, depression-dejection, vigor-activity, fatigue-inertia, and confusion-bewilderment. Adjectives are rated on a scale 1 (not at all) to 6 (extremely).
Measure latency to sleep using the Maintenance of Wakefulness Test (MWT) | Performed at approximately 75 minute intervals (+/-10 minutes) throughout the waking period, beginning approximately one hour post-awakening on the day prior to sleep restriction and on the recovery day and on the night of sleep restriction. Days 11 - 15
  Subjects will be escorted to their individual darkened, sound-attenuated bedrooms and allowed to lie down on their beds. They will be instructed to close their eyes and try to remain awake. Polysomnography will be monitored online.
Measure alertness using the Karolinska Sleepiness Scale (KSS) | Performed at approximately 75 minute intervals (+/-10 minutes) throughout the waking period, beginning approximately one hour post-awakening on the day prior to sleep restriction and on the recovery day and on the night of sleep restriction. Days 11 - 15
  Computer based self rated level of alertness ranging from 1 (extremely alert to 9 (extremely sleepy).
Measure of declarative or associative learning using the Paired Word Associates Task (PWAT) | Within 60 minutes of bedtime on the sleep restriction night with a recall phase conducted approximately 20 and 120 minutes after awakening on the same night. Days 11 and 12
  46 word pairs will be administered in a learning phase. Four additional word pairs will be administered at the beginning and end of the 46 pair test list during the learning phase in order to minimize primacy and recency learning effects, but will not be part of the recall phase.

CONTACTS AND LOCATIONS:
Overall Officials: John D. Hughes, CDR, MC, USN, Principal Investigator — Naval Medical Research Center
Locations (1):
- Naval Medcical Research Center (NMRC) Clincal Trials Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No